CLINICAL TRIAL: NCT02147145
Title: Prospective Database of Gastrointestinal Stromal Cell Tumors (GISTs)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: ProGIST 1
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Gastrointestinal Stromal Cell Tumors; Foregut Subepithelial Lesions
Keywords: GIST; endoscopy; endoscopic ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years

GROUPS / COHORTS (1):
- Observation Cohort

SUMMARY:
Specific Aim 1: To determine patient compliance with a GIST surveillance program Hypothesis: Patient compliance with a GIST surveillance program will be low.

Specific Aim 2: To determine if EUS features of GIST, particularly maximum size, change significantly during a surveillance program.

Hypothesis: EUS features of GIST, particularly maximum size, will not change significantly during a surveillance program.

Specific Aim 3: To determine if EGD measures of GIST size correlate well with EUS measures of GIST size.

Hypothesis: EGD measures of GIST size will correlate well with EUS measured of GIST size.

ELIGIBILITY:
Inclusion Criteria:

* presenting for EUS with an indication for a SEL in the stomach or esophagus
* at least 18 years of age
* able to provide informed consent

Exclusion Criteria:

* no subepithelial lesion in the stomach or esophagus'
* less than 18 years of age
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years of age) referred for EUS evaluation of incidentally discovered foregut SEL at a two tertiary care centers between 8/2008 and 8/2012.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Determine the natural history of small (< 30 mm) SELs discovered evaluated by EUS. | 3 years

SECONDARY OUTCOMES:
Determine the degree of patient compliance with surveillance recommendations. | 3 years
Describe the diagnostic yield of EUS±FNA in evaluating SELs. | 2 weeks
Compare SEL size estimation based on EUS, EGD and computer tomography (CT). | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States